CLINICAL TRIAL: NCT01155011
Title: MIPARC - Multilevel Intervention for Physical Activity in Retirement Communities
Brief Title: Multilevel Intervention for Physical Activity in Retirement Communities
Acronym: MIPARC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Jacqueline Kerr, Assistant Professor, Department of Family and Preventive Medicine, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 3134795; 1R01HL098425 (NIH)
Record Dates: First submitted 2010-06-30; First posted 2010-07-01 (Estimated); Results first posted 2017-07-31 (Actual); Last update posted 2017-08-31 (Actual); Status verified 2017-08

CONDITIONS: Physical Activity; Blood Pressure; Physical Functioning; Quality of Life; Sedentary
Keywords: Older adults; physical activity; sedentary; retirement communities; advocacy; built environment; peer mentoring; walkability
MeSH Terms: conditions — Motor Activity; Sedentary Behavior | interventions — Exercise; Palliative Care

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MIPARC intervention (Experimental): Eleven Continuing Care Retirement Communities were randomized to either the MIPARC intervention or an attention-control condition. The intervention focused on increasing light to moderate PA.
  The MIPARC study intervenes on four levels: individual (pedometer self monitoring, educational materials and monthly counseling calls, support), interpersonal (monthly group educational sessions and peer mentoring), environment (walking signage prompts, tailored environmental resources, step counts)and policies (review of on-site activity opportunities and walkability, recommendations for policy change and peer led advocacy)to increase the activity levels of residents.
  For the first 3 months, intervention participants will engage in either a group educational session, phone counseling call, or a peer led session, on a rotating basis.
  Interventions: Behavioral: Physical Activity; Behavioral: Group educational sessions; Behavioral: Phone counseling call; Behavioral: Peer Mentoring; Behavioral: Policy Change; Behavioral: Support; Behavioral: Tailored environmental resources
- Health Education Control (Active Comparator): The control group received an active health education intervention. The education curriculum will involve both lectures and mailed materials. The lectures were delivered to match the MIPARC intervention schedule. Sessions included information on general health and healthy aging. Physical activity was not discussed in these sessions but participants received information on the benefits of PA. Control participants also received health check phone calls to match the individual attention paid to participants in the MIPARC intervention sites.
  Interventions: Behavioral: Group educational sessions; Behavioral: Health check phone call; Behavioral: Pedometer

INTERVENTIONS:
Behavioral: Physical Activity — MIPARC will focus on 3 physical activity goals:
  1. increasing walking behavior through gradually increasing step goals
  2. increasing attendance at available on-site and local aerobic, strength and flexibility classes, as well as prompting stair use,
  3. reducing sedentary behavior. Participants will monitor their steps with a pedometer, daily step logs and progress charts. All participants will have a gradually increasing fixed step goal for each week that will result in an total increase of 3000 steps after 3 months, which they will be supported to maintain for an additional 3 months.
  Arms: MIPARC intervention
Behavioral: Group educational sessions — Every three weeks, participants will be required to attend a group education session, where researchers will teach behavior change strategies and allow participants to share their experiences and offer support to each other. The group sessions will follow a common format including: a group exercise (e.g. quiz), group discussion of use of behavior change strategies (e.g. overcoming barriers), and will end with a behavior change strategy instruction and goal setting component.
  Arms: MIPARC intervention
Behavioral: Phone counseling call — To support a tailored intervention delivery, participants will receive 4 individual phone calls (in weeks 2, 5, 8, and 11) from a trained health counselor. The phone call will follow the following format:
  1. health check
  2. step goal check
  3. barrier identification
  4. problem solving
  5. specific goals to achieve target step counts. Counselors will prompt participants to report any adverse events, illnesses, medication changes or counter indicative symptoms. The calls will cease during the second 3 months to allow participants to practice self help techniques while still supported by the group sessions and peer mentoring.
  Arms: MIPARC intervention
Behavioral: Peer Mentoring — Three peer mentors at each CCRC will be trained in intervention content and delivery, measurement support, and advocacy. The peer mentors will lead a group session once every three weeks for the 6 month intervention period and once a month for the following 6 months. The peer mentors will formulate their own ideas for these sessions but we will suggest they include group walks, group activities and trips to active locations, etc.
  The peers will help study staff to answer questions from participants and assist with study compliance and retention. They will also receive advocacy training from a non-profit advocacy organization to conduct walk audits of their CCRC and help mobilize participants to make changes to their community that will increase or improve the opportunities for physical activity.
  Arms: MIPARC intervention
Behavioral: Policy Change — In order to increase the sustainability of the project, MIPARC will focus on addressing on-site policies and neighborhood factors that are barriers to physical activity. Peers and staff will conduct site inspections to identify these barriers (e.g. lack of facilities, limited opening hours, unsafe sidewalks, etc.) which will be prioritized and presented to CCRC management and community officials.
  Arms: MIPARC intervention
Behavioral: Support — A binder of professionally prepared materials will be provided at the beginning of the intervention and are referred to by researchers in the group sessions and phone counseling calls. The materials provide important information to encourage knowledge, self efficacy and realistic expectations.
  Arms: MIPARC intervention
Behavioral: Tailored environmental resources — Participants will be provided with a set of printed materials relating to the residential and neighborhood environment of their CCRC. A list of step counts for key indoor routes will be provided as well as safe walking route maps for the site an local neighborhood.
  Arms: MIPARC intervention
Behavioral: Group educational sessions — Lectures will be delivered every three weeks to match the MIPARC intervention schedule. Sessions will include topics such as medications, foot care and nutrition. Physical activity will not e discussed in these sessions but participants will receive informational pamphlets on the benefits of physical activity.
  Arms: Health Education Control
Behavioral: Health check phone call — For the first 3 months, control participants will also receive a health check phone call to match the individual attention paid to participants in the MIPARC sites.
  Arms: Health Education Control
Behavioral: Pedometer — Participants will also keep the pedometer they wear during the baseline measurement week to satisfy any curiosity about the devices and the step entry criteria. They will be given instructions on its use but will not be taught the benefits of self-monitoring.
  Arms: Health Education Control

SUMMARY:
The purpose of this study was to assess whether a 6-month multilevel physical activity intervention can significantly increase physical activity levels in sedentary adults, 65 and older, living in Continuing Care Retirement Communities (CCRCs).

Sedentary residents (N=307) in 11 CCRCs received the multilevel MIPARC intervention or a control health education program for 6 months. A group randomized control design was employed with site as the unit of randomization. The intervention was delivered through group sessions, phone calls, printed materials, tailored signage and mapping and targeted peer led advocacy efforts.

DETAILED DESCRIPTION:
Objective monitoring of physical activity suggests that fewer than 3% of adults over age 60 meet current physical activity guidelines. Ecological models posit that behavioral interventions are most effective when they operate on multiple levels. The MIPARC study intervenes on four levels: individual (pedometer-based self monitoring, educational materials and monthly counseling calls), interpersonal (monthly group sessions and peer mentoring), environment (walking signage prompts, tailored walking maps, step counts)and policies (review of on-site activity opportunities and walkability, recommendations for change and peer led advocacy)to increase the activity levels of residents. The study promotes walking as the primary means to increase light to moderate PA, with a secondary focus on strength and flexibility and decreased sedentary behavior.

As most Continuing Care Retirement Communities have management structures that provide the opportunity to improve the social and built environments for physical activity and walking, this study also aims to train participants on how to advocate for improvements in the environment that would improve walkability.

ELIGIBILITY:
Inclusion Criteria:

* Over the age of 65
* Able to walk 20 meters independently (without human assistance, can use cane/walker)
* Able to speak and read in English
* No cognitive, vision or hearing impairments that would prevent provision of informed consent, comprehension of instructions, completion of surveys and participation in phone conversations
* Able to complete the Timed Up and Go Test to assess falls risk within 30 seconds
* Live within the selected retirement community (facility-dwelling) Able to hold brief conversation over the telephone.
* Will be in San Diego for the duration of the study
* Provision of consent to participate
* Willing to wear a pedometer, accelerometer and GPS device
* Willing to complete all surveys and attend weekly meetings
* No history of falls in previous that resulted in an injury or hospitalization in the past 12 months
* Physician clearance to participate

Exclusion Criteria:

* Inability to give informed, voluntary consent
* Inability to complete assessments
* Lack of written physician consent to participate in unsupervised light-to-moderate intensity walking
* Inability to speak and read English

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 307 (Actual)
Dates: Start 2011-01; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline Kerr, PhD, Principal Investigator — University of California, San Diego
Locations (1):
- University of California, San Diego, La Jolla, California, United States

REFERENCES:
- [Background] Rosenberg D, Kerr J, Sallis JF, Patrick K, Moore DJ, King A. Feasibility and outcomes of a multilevel place-based walking intervention for seniors: a pilot study. Health Place. 2009 Mar;15(1):173-9. doi: 10.1016/j.healthplace.2008.03.010. Epub 2008 Apr 8. PMID 18502164
- [Background] Kerr J, Rosenberg DE, Nathan A, Millstein RA, Carlson JA, Crist K, Wasilenko K, Bolling K, Castro CM, Buchner DM, Marshall SJ. Applying the ecological model of behavior change to a physical activity trial in retirement communities: description of the study protocol. Contemp Clin Trials. 2012 Nov;33(6):1180-8. doi: 10.1016/j.cct.2012.08.005. Epub 2012 Aug 17. PMID 22921641
- [Background] Bellettiere J, Carlson JA, Rosenberg D, Singhania A, Natarajan L, Berardi V, LaCroix AZ, Sears DD, Moran K, Crist K, Kerr J. Gender and Age Differences in Hourly and Daily Patterns of Sedentary Time in Older Adults Living in Retirement Communities. PLoS One. 2015 Aug 21;10(8):e0136161. doi: 10.1371/journal.pone.0136161. eCollection 2015. PMID 26296095
- [Background] Kerr J, Marshall SJ, Patterson RE, Marinac CR, Natarajan L, Rosenberg D, Wasilenko K, Crist K. Objectively measured physical activity is related to cognitive function in older adults. J Am Geriatr Soc. 2013 Nov;61(11):1927-31. doi: 10.1111/jgs.12524. PMID 24219194
- [Background] Marshall S, Kerr J, Carlson J, Cadmus-Bertram L, Patterson R, Wasilenko K, Crist K, Rosenberg D, Natarajan L. Patterns of Weekday and Weekend Sedentary Behavior Among Older Adults. J Aging Phys Act. 2015 Oct;23(4):534-41. doi: 10.1123/japa.2013-0208. Epub 2014 Nov 21. PMID 25415205
- [Background] Rosenberg DE, Bellettiere J, Gardiner PA, Villarreal VN, Crist K, Kerr J. Independent Associations Between Sedentary Behaviors and Mental, Cognitive, Physical, and Functional Health Among Older Adults in Retirement Communities. J Gerontol A Biol Sci Med Sci. 2016 Jan;71(1):78-83. doi: 10.1093/gerona/glv103. Epub 2015 Aug 13. PMID 26273024
- [Result] Takemoto M, Carlson JA, Moran K, Godbole S, Crist K, Kerr J. Relationship between Objectively Measured Transportation Behaviors and Health Characteristics in Older Adults. Int J Environ Res Public Health. 2015 Oct 30;12(11):13923-37. doi: 10.3390/ijerph121113923. PMID 26528999
- [Derived] Kerr J, Rosenberg D, Millstein RA, Bolling K, Crist K, Takemoto M, Godbole S, Moran K, Natarajan L, Castro-Sweet C, Buchner D. Cluster randomized controlled trial of a multilevel physical activity intervention for older adults. Int J Behav Nutr Phys Act. 2018 Apr 2;15(1):32. doi: 10.1186/s12966-018-0658-4. PMID 29609594

RESULTS

PARTICIPANT FLOW:
Groups:
- MIPARC Intervention: The intervention will focus on increasing light to moderate PA, primarily promoting walking by gradually increasing participants' daily step counts.
  Participants will monitor their steps with a pedometer, daily step logs and progress charts. All participants will have a gradually increasing fixed step goal for each week that will result in an total increase of 3000 steps after 3 months, which they will be supported to maintain for an additional 3 months. Participants will attend group educational sessions and group walks, receive phone counseling calls from UCSD counselors, receive support from peer mentors, In order to increase the sustainability of the project, MIPARC will focus on addressing on-site policies and neighborhood factors that are barriers to physical activity.
- Health Education Control: The control group will receive an active health education intervention. The education curriculum will involve both lectures and mailed materials. The lectures will be delivered to match the MIPARC intervention schedule. Sessions will include information on general health and healthy aging. Physical activity will not be discussed in these sessions but participants will receive information on the benefits of PA. Control participants will also receive a health check phone call to match the individual attention paid to participants in the MIPARC intervention sites.
Period: Baseline to 6 Months
Arm/Group | MIPARC Intervention | Health Education Control
Started | 151 | 156
Completed | 129 | 131
Not Completed | 22 | 25
Not completed — Withdrawal by Subject | 18 | 19
Not completed — investigator decision, moved | 4 | 5
Not completed — Death | 0 | 1
Period: 6 to 12 Months
Arm/Group | MIPARC Intervention | Health Education Control
Started | 129 | 131
Completed | 120 | 121
Not Completed | 9 | 10
Not completed — Withdrawal by Subject | 8 | 5
Not completed — Death | 1 | 5

BASELINE CHARACTERISTICS:
Groups:
- MIPARC Intervention: Intervention participants engage in group education session, individual phone counseling calls and group walks for the first 6 months. The telephone counseling calls will be eliminated after 3 months.
  Participants monitor their steps with a pedometer, daily step logs and progress charts. All participants will have a gradually increasing fixed step goal for each week that will result in an total increase of 3000 steps after 3 months, which they will be supported to maintain for an additional 3 months. They receive support from peer leaders. The peer leaders also receive advocacy training from a non-profit advocacy organization to conduct walk audits of their CCRC and help mobilize participants to make changes to their community that will increase or improve the opportunities for physical activity.
- Health Education Control: The control group will receive an active health education intervention. The lectures will be delivered to match the MIPARC intervention schedule. Sessions will include information on general health and healthy aging. Physical activity will not be discussed in these sessions but participants will receive information on the benefits of PA. Control participants will also receive a health check phone call to match the individual attention paid to participants in the MIPARC intervention sites.
- Total: Total of all reporting groups
Arm/Group | MIPARC Intervention | Health Education Control | Total
Number analyzed (Participants) | 151 | 156 | 307
Age, Continuous [Mean (Standard Deviation); unit: years] | 85.3 (6.5) | 81.9 (5.9) | 83.6 (6.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 107 | 115 | 222
  Male | 44 | 41 | 85
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 4
  Not Hispanic or Latino | 148 | 151 | 299
  Unknown or Not Reported | 2 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 3
  Asian | 14 | 1 | 15
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 132 | 150 | 282
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 0 | 3 | 3
Education [Number; unit: participants] — College education and above
  participants | 91 | 108 | 199
Marital Status [Count of Participants; unit: Participants] — Married
  Participants | 45 | 81 | 126

OUTCOME MEASURES:

1. Primary Outcome: Daily Minutes of Physical Activity
Description: Measured by 7 day accelerometry with a 760 cpm cutpoint.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- MIPARC Intervention: Intervention participants received group education sessions, group walks, phone counseling and support from peer leaders.
- Health Education Control: The control group will receive an active health education intervention. The lectures will be delivered to match the MIPARC intervention schedule. Sessions will include information on general health and healthy aging. Physical activity will not be discussed in these sessions but participants will receive information on the benefits of PA.
Arm/Group | MIPARC Intervention | Health Education Control
Number analyzed (Participants) | 151 | 156
minutes | 50.03 (29.02) | 39.19 (28.3)

2. Primary Outcome: Daily Minutes of Physical Activity
Description: Measured by 7 day accelerometry in adults, ≥65, with a 760 CPM cutpoint.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- MIPARC Intervention: Participants received group educations sessions, group walks, phone counseling, support from peer leaders.
- Health Education Control: The control group will receive an active health education intervention.. The lectures will be delivered to match the MIPARC intervention schedule.
Arm/Group | MIPARC Intervention | Health Education Control
Number analyzed (Participants) | 124 | 127
minutes | 59.46 (40.05) | 39.24 (25.11)

3. Primary Outcome: Minutes of Light to Moderate Physical Activity
Description: Measured by 7 day accelerometry in adults, ≥65, using a 760 CPM cutpoint.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- MIPARC Intervention: Intervention participants engage in group education session, individual phone counseling calls and group walks for the first 6 months. The telephone counseling calls will be eliminated after 3 months.
  Participants monitor their steps with a pedometer, daily step logs and progress charts. All participants will have a gradually increasing fixed step goal for each week that will result in an total increase of 3000 steps after 3 months, which they will be supported to maintain for an additional 3 months. They receive support from peer leaders.
Arm/Group | MIPARC Intervention | Health Education Control
Number analyzed (Participants) | 110 | 107
minutes | 56.79 (38.32) | 38.70 (26.50)

ADVERSE EVENTS:
Arm/Group | MIPARC Intervention | Health Education Control
All-Cause Mortality (participants affected / at risk) | 1/151 | 5/156
Serious Adverse Events (participants affected / at risk) | 38/151 | 30/156
Other Adverse Events (participants affected / at risk) | 23/151 | 12/156
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MIPARC Intervention (N=151) | Health Education Control (N=156)
Death (General disorders) | 1 (1) | 5 (5)
Fall (General disorders) | 20 (20) | 16 (16)
Serious physical injury (Musculoskeletal and connective tissue disorders) | 5 (5) | 1 (1)
Persistent or significant physical or cognitive disability or incapacity (General disorders) | 3 (3) | 3 (3)
Overnight hospitalization (General disorders) | 10 (10) | 5 (5) — Any reason
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MIPARC Intervention (N=151) | Health Education Control (N=156)
Change in care status (General disorders) | 1 (1) | 0 (0)
Emergency room visit (General disorders) | 3 (3) | 3 (3)
Other (General disorders) | 19 (19) | 8 (8) — reported pain, arthritis, autoimmune disorder or infections
Decreased cognition (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No